CLINICAL TRIAL: NCT03758924
Title: A Double-Blind, Randomized, Placebo-Controlled, Dose Titration Study of ANAVEX2-73 in Patients With Rett Syndrome
Brief Title: Study of ANAVEX2-73 in Patients With Rett Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anavex Life Sciences Corp. (Industry)
Collaborators: International Rett Syndrome Foundation Rettsyndrome.org (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANAVEX2-73-RS-001
Record Dates: First submitted 2018-11-25; First posted 2018-11-29 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Rett Syndrome
MeSH Terms: conditions — Rett Syndrome | interventions — tetrahydro-N, N-dimethyl-2,2-diphenyl-3-furanmethanamine hydrochloride

STUDY DESIGN:
Intervention Model Description: 31 participants: 6 PK open-label followed by 25 double-blind, randomized, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind, Randomized, Placebo-Controlled
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active arm (Experimental): Week 0-7: Take 1 ml orally of the product daily (solution of ANAVEX2-73)
  Interventions: Drug: ANAVEX2-73
- Placebo arm (Placebo Comparator): Week 0-7: Take 1 ml orally of the product daily (placebo)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ANAVEX2-73 — Liquid oral solution
  Arms: Active arm
Drug: Placebo — Liquid oral solution
  Arms: Placebo arm

SUMMARY:
Phase 2 safety, tolerability and efficacy study is designed as a double-blind, randomized, placebo-controlled study.

7-week placebo-controlled study of ANAVEX2-73 oral solution for the treatment of patients with RTT 18 years or older. A voluntary option will be offered for all patients who meet the exposure criteria for ANAVEX2-73 to continue a 12-week open label extension.

DETAILED DESCRIPTION:
This Phase 2 safety, tolerability and efficacy study is designed as a double-blind, randomized, placebo-controlled study.

This is a 7-week placebo-controlled study of ANAVEX2-73 oral solution for the treatment of patients with RTT 18 years or older. A voluntary option will be offered for all patients who meet the exposure criteria for ANAVEX2-73 to continue a 12-week open label extension.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years, inclusive.
* Diagnosis of classic RTT, according to 2010 criteria (Neul et al., 2010), and a MECP2 mutation.
* Current pharmacological treatment regimen, including supplements, has been stable for at least 4 weeks.
* If on antiepileptic drugs (AEDs), 1-4 AEDs allowed. Treatment must be stable (drug, dose, interval of administration) for 30 days prior to enrollment.
* Ability to keep accurate seizure diaries or have caregiver who can keep accurate seizure diaries.
* Confirmation from the participant that, if of childbearing potential is not pregnant through urine pregnancy testing. Female patients of childbearing potential and at risk for pregnancy must agree to abstinence.
* Prior to the conduct of study-specific procedures, the subject's parent/caregiver/LAR must provide written informed consent. If applicable, the research team must attempt to obtain consent from both parents.

Exclusion Criteria:

* Patients who have a progressive medical or neurological condition that in the opinion of the Investigator would interfere with the conduct of the study.
* Current clinically significant systemic illness that is likely to result in deterioration of the patient's condition or affect the patient's safety during the study.
* History of clinically evident stroke or clinically significant carotid or vertebrobasilar stenosis or plaque or other history of neurologic (e.g., head trauma with loss of consciousness) or psychiatric condition that the Investigator deems may interfere with interpretability of data.
* Indication of liver disease, defined by serum levels of ALT (SGPT), AST (SGOT), or alkaline phosphatase above 3x upper limit of normal (ULN) as determined during screening.
* Treatment with immunosuppressive medications (e.g., systemic corticosteroids) within the last 90 days (topical and nasal corticosteroids and inhaled corticosteroids for asthma are permitted) or chemotherapeutic agents for malignancy within the last 3 years.
* Other clinically significant abnormality on physical, neurological, laboratory, or electrocardiogram (ECG) examination (e.g., atrial fibrillation) that could compromise the study or be detrimental to the participant.
* Any known hypersensitivity to any of the excipients contained in the study drug or placebo formulation.
* Other co-morbid or chronic illness beyond that known to be associated with RTT.
* Subjects who plan to initiate or change pharmacologic or nonpharmacologic intervention during the course of the study.
* Subjects on potent CYP 3A4 and CYP2C19 inhibitors and inducers.
* Subjects taking another investigational drug currently or within the last 30 days.
* Any other criteria (such as a clinically significant screening blood test result), which in the opinion of the Investigator could interfere with the study conduct or outcome.
* Patients with hepatic and renal impairment.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events | 7 weeks
  Incidence of Adverse Events
Maximum Plasma Concentration [Cmax] of ANAVEX2-73 | 7 weeks
  PK of ANAVEX2-73 and metabolite
Area Under the Curve [AUC] of ANAVEX2-73 | 7 weeks
  PK of ANAVEX2-73 and metabolite
Lipid panel | 7 weeks
  Significant laboratory findings

SECONDARY OUTCOMES:
RSBQ | 7 weeks
  Change from baseline to End of Treatment (EOT) in the Rett Syndrome Behaviour Questionnaire (RSBQ). Total score and a pre-specified subset of the RSBQ
CGI-I | 7 weeks
  Change from baseline to End of Treatment (EOT) in the Clinical Global Impression Improvement Scale (CGI-I) score. Total score and a pre-specified subset of the CGI-I

OTHER OUTCOMES:
Anxiety, Depression, and Mood Scale (ADAMS) | 7 weeks
  Anxiety, Depression, and Mood Scale (ADAMS)
Children's Sleep Habits Questionnaire (CSHQ) | 7 weeks
  Children's Sleep Habits Questionnaire (CSHQ)
Visual Analog Scale (VAS) | 7 weeks
  Visual Analog Scale (VAS)
Seizure Frequency via seizure diary | 7 weeks
  Seizure Frequency via seizure diary
Genetic variant SIGMAR1, COMT | 7 weeks
  Pre-specified endpoint
Glutamate Plasma Concentration | 7 weeks
  Biomarker
GABA Plasma Concentration | 7 weeks
  Biomarker

CONTACTS AND LOCATIONS:
Overall Officials: Walter Kaufmann, MD, Principal Investigator — Emory University SOM
Locations (8):
- United States (8):
  - UAB | The University of Alabama at Birmingham, Birmingham, Alabama
  - UC Davis University of California - Davis MIND Institute, Sacramento, California
  - Rush University Medical Center, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Washington University in St. Louis | Saint Louis Children's Hospital, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Greenwood Genetic Center, Greenwood, South Carolina
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No